CLINICAL TRIAL: NCT02306148
Title: Effects of a Foot Strengthening Program on the Incidence of Injuries, Foot Functionality and Health in Long Distance Runners: a Randomized Controlled Trial.
Brief Title: Effects of Foot Strengthening on the Incidence of Injuries in Long Distance Runners
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sao Paulo General Hospital (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado de São Paulo (Other Government)
Responsible Party: Principal Investigator, Isabel de Camargo Neves Sacco, Associate Professor, University of Sao Paulo General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: LaBiMPH-002
Record Dates: First submitted 2014-11-28; First posted 2014-12-03 (Estimated); Results first posted 2024-05-28 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2023-12

CONDITIONS: Leg Injuries
MeSH Terms: conditions — Leg Injuries

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Group (Placebo Comparator): Group will practice 15 seconds isometric lower limb stretching protocol and must continue practicing running as usual.
  Interventions: Other: Foot and ankle strengthening
- Foot and ankle strengthening (Experimental): Group will be trained during 2 months by a physiotherapist for foot and ankle strengthening and must continue to exercise at home with a training software supervision. Must continue practicing running as usual.
  Interventions: Other: Foot and ankle strengthening

INTERVENTIONS:
Other: Foot and ankle strengthening — Group will be trained during 2 months at the university by a physiotherapist and at home with a training software for foot and ankle strengthening.

SUMMARY:
The main objective of this trial is to investigate the effects of a training protocol for the foot and ankle complex on the prevalence of running related injuries on long distance runners.

DETAILED DESCRIPTION:
Using a web software as a follow up tool, subjects can be scanned for injuries and have them confirmed by a physician, determining the injuries prevalence in one year.

Through force platform and infrared cameras, the kinematics and kinetics during gait will allow assessment of joint moments, power during propulsion, ankle and knee range of motion.

The hypothesis is that a strengthening program for foot and ankle muscles can alter the prevalence of lower limbs injuries on long distance runners, lowering the harmful forces that these segments receive. The participants will be randomly assigned into control group (placebo intervention) or into intervention group, that will receive an 8 weeks strengthening intervention, twice a week with the supervision of a physiotherapist and three times a week being remotely supervised by a software at home, for 30 minutes each session. This will aim for increasing foot and ankle range of movement and muscle strength.

Every exercise has its own progression depending on the subjects execution, increasing in intensity and difficulty.

ELIGIBILITY:
Inclusion Criteria:

* practice long distance (more than 5 km) running for at least one year;
* run at least 20 km a week;

Exclusion Criteria:

* run using minimalist shoes or barefoot;
* having prior experience in isolated foot and ankle strength training within the last year;
* have any health condition that affect gait and running;
* being receiving any physical therapy intervention;
* having any running related injuries during the last two months.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 118 (Actual)
Dates: Start 2015-04; Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Isabel Sacco, PHD, Principal Investigator — Associate Professor at São Paulo University
Locations (1):
- Universidade de São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
All files are available in the database published at http://figshare.com after completion of the study. All metadata are also available at m https://repositorio.uspdigital.usp.br/
Time Frame: after completion of the study.
Access Criteria: Upon request.
URL: https://doi.org/10.6084/m9.figshare.10003406.v1

REFERENCES:
- [Derived] Suda EY, Watari R, Matias AB, Taddei UT, Sacco ICN. Predictive Effect of Well-Known Risk Factors and Foot-Core Training in Lower Limb Running-Related Injuries in Recreational Runners: A Secondary Analysis of a Randomized Controlled Trial. Am J Sports Med. 2022 Jan;50(1):248-254. doi: 10.1177/03635465211056329. Epub 2021 Nov 17. PMID 34786990
- [Derived] Watari R, Suda EY, Santos JPS, Matias AB, Taddei UT, Sacco ICN. Subgroups of Foot-Ankle Movement Patterns Can Influence the Responsiveness to a Foot-Core Exercise Program: A Hierarchical Cluster Analysis. Front Bioeng Biotechnol. 2021 Jun 8;9:645710. doi: 10.3389/fbioe.2021.645710. eCollection 2021. PMID 34169063
- [Derived] Taddei UT, Matias AB, Duarte M, Sacco ICN. Foot Core Training to Prevent Running-Related Injuries: A Survival Analysis of a Single-Blind, Randomized Controlled Trial. Am J Sports Med. 2020 Dec;48(14):3610-3619. doi: 10.1177/0363546520969205. Epub 2020 Nov 6. PMID 33156692
- [Derived] Matias AB, Taddei UT, Duarte M, Sacco IC. Protocol for evaluating the effects of a therapeutic foot exercise program on injury incidence, foot functionality and biomechanics in long-distance runners: a randomized controlled trial. BMC Musculoskelet Disord. 2016 Apr 14;17:160. doi: 10.1186/s12891-016-1016-9. PMID 27075480
- See also: Laboratory website — http://www.usp.br/labimph
- See also: University website — http://www.fm.usp.br/

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control Group | Foot and Ankle Strengthening
Started | 61 | 57
Completed | 48 | 47
Not Completed | 13 | 10
Not completed — Adverse Event | 12 | 6
Not completed — Lost to Follow-up | 1 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | Foot and Ankle Strengthening | Total
Number analyzed (Participants) | 61 | 57 | 118
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 61 | 57 | 118
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.3 (6.85) | 40.5 (7.9) | 40.9 (7.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29 | 29 | 58
  Male | 32 | 28 | 60
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Brazil | 61 | 57 | 118
Running experience (years) [Mean (Standard Deviation); unit: years] | 6.9 (5.8) | 5.4 (4.7) | 6.2 (5.3)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Running Related Lower Limb Injuries
Description: Diagnosed running related lower limb injuries in recreational runners within 12 months of the study
Time Frame: 1 year
Measure: Count of Participants; unit: Participants
Arm/Group | Control Group | Foot and Ankle Strengthening
Number analyzed (Participants) | 61 | 57
Participants | 20 | 8

2. Secondary Outcome: Time to the First Injury
Description: How long it takes to a diagnosed running related lower limb injuries to occur
Time Frame: 12 months
Population: 25% quartile-estimation of time-to-injury survival time
Measure: Mean (Standard Deviation); unit: months
Arm/Group | Control Group | Foot and Ankle Strengthening
Number analyzed (Participants) | 61 | 57
months | 10.15 (2.69) | 7.63 (2.60)

3. Secondary Outcome: Toes and Hallux Muscle Strength
Description: Outcome measure under the hallux summed to toes while the subject is pressing their toes against a pressure sensor platform (sum of toes and hallux strength)
Time Frame: 2 months
Population: 2x2 repeated measures analysis of variance (ANOVA) was used to compare the interaction effect of training (foot strengthening vs. control) and time (T0 and T8). In case of significant interaction effects, Tukey's HSD test was used to conduct pairwise comparisons to identify differences in time, group, or both.
Measure: Mean (Standard Deviation); unit: %bodyweight
Arm/Group | Control Group | Foot and Ankle Strengthening
Number analyzed (Participants) | 61 | 57
%bodyweight | 25.61 (7.40) | 27.31 (9.33)

4. Secondary Outcome: Foot Muscles Hypertrophy (Volume)
Description: Intrinsic foot muscles volume measured by MRI
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: cm3
Arm/Group | Control Group | Foot and Ankle Strengthening
Number analyzed (Participants) | 14 | 14
cm3
  Abductor Hallucis volume | 13.3 (6.3) | 13.7 (6.3)
  flexor digitorum brevis volume | 13.3 (4.3) | 12.5 (4.7)
  abductor digiti minimi volume | 12.0 (4.6) | 11.2 (4.8)
  flexor hallucis brevis volume | 12.0 (4.1) | 10.2 (4.4)

5. Secondary Outcome: Foot Health and Functionality
Description: Score of the Foot Health Status questionnaire - Brazilian version (domains: function and general foor health) - Scale of FHSQ (0-100 max, the higher the better)
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Control Group | Foot and Ankle Strengthening
Number analyzed (Participants) | 61 | 57
units on a scale
  General Foot health | 83 (27.6) | 92 (11.6)
  Foot function | 100 (0.0) | 100 (1.7)

6. Secondary Outcome: Foot and Ankle Running Kinematics
Description: medial longitudinal arch range of motion during barefoot running on a treadmill
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Control Group | Foot and Ankle Strengthening
Number analyzed (Participants) | 61 | 57
degrees | 2.88 (5.36) | 0.17 (6.86)

7. Secondary Outcome: Ground Reaction Forces During Running
Description: Breaking forces (negative values as it is a decceleration force), vertical peak forces (positive values) measured on a force platform during subject's runnning
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: *bodyweight
Arm/Group | Control Group | Foot and Ankle Strengthening
Number analyzed (Participants) | 41 | 46
*bodyweight
  Vertical force peak (BW) | 1.09 (0.58) | 1.14 (0.55)
  Peak Breaking force (BW) (negative values as it is a decceleration force) | -0.24 (0.05) | -0.24 (0.07)

8. Secondary Outcome: Foot Inversion During Running
Description: Shank to calcaneous inversion angle during barefoot running on a treadmill
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Control Group | Foot and Ankle Strengthening
Number analyzed (Participants) | 41 | 46
degrees | -3.51 (5.7) | -5.74 (6.31)

9. Secondary Outcome: Foot Eversion During Running
Description: Shank to calcaneous eversion angle during barefoot running on a treadmill
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: degrees
Arm/Group | Control Group | Foot and Ankle Strengthening
Number analyzed (Participants) | 41 | 46
degrees | 6.39 (1.88) | 5.90 (2.95)

10. Secondary Outcome: Vertical Loading Rate Force During Running
Description: Vertical loading rate measured on a force platform during subject's runnning
Time Frame: 2 months
Measure: Mean (Standard Deviation); unit: *bodyweight/s
Arm/Group | Control Group | Foot and Ankle Strengthening
Number analyzed (Participants) | 41 | 46
*bodyweight/s | 72.84 (65.73) | 77.17 (57.52)

ADVERSE EVENTS:
Time Frame: 1 year
Description: Adverse Events was defined as in clinicaltrials.gov
Arm/Group | Control Group | Foot and Ankle Strengthening
All-Cause Mortality (participants affected / at risk) | 0/61 | 0/57
Serious Adverse Events (participants affected / at risk) | 0/61 | 0/57
Other Adverse Events (participants affected / at risk) | 0/61 | 0/57

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2016-05-01): https://cdn.clinicaltrials.gov/large-docs/48/NCT02306148/Prot_SAP_000.pdf
  • Informed Consent Form (2015-03-01): https://cdn.clinicaltrials.gov/large-docs/48/NCT02306148/ICF_001.pdf